CLINICAL TRIAL: NCT07053566
Title: Effects of Latissimus Dorsi Exercises on Acromiohumeral Interval, Pain, and Function in Rotator Cuff Tendinopathy
Brief Title: Latissimus Dorsi Strengthening Exercises in Rotator Cuff Tendinopathy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Irem Duzgun, Professor and Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LDRCT
Record Dates: First submitted 2025-06-18; First posted 2025-07-08 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-06

CONDITIONS: Rotator Cuff Related Shoulder Pain; Rotator Cuff Tendinopathy; Subacromial Impingement Syndrome
Keywords: Exercise Theraphy; Shoulder Rehabilitation; Rotator Cuff; Latissimus Dorsi
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Investigator
Masking Description: In this study, both the participants and the investigator (physician) are blinded to the group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Rotator Cuff Exercise Group (RCEG) (Experimental): Progressive strengthening program for rotator cuff muscles.
  Interventions: Behavioral: Rotator Cuff Strengthening Exercises
- Latissimus Dorsi Exercise Group (LDEG) (Experimental): Progressive strengthening program for latissimus dorsi muscle.
  Interventions: Behavioral: Latissimus Dorsi Strengthening Exercises
- Combined Exercise Group (CEG) (Experimental): Combined strengthening program for rotator cuff and latissimus dorsi muscles
  Interventions: Behavioral: Rotator Cuff Strengthening Exercises; Behavioral: Latissimus Dorsi Strengthening Exercises

INTERVENTIONS:
Behavioral: Rotator Cuff Strengthening Exercises — Progressive exercise program focused on rotator cuff muscles
  Arms: Combined Exercise Group (CEG); Rotator Cuff Exercise Group (RCEG)
Behavioral: Latissimus Dorsi Strengthening Exercises — Progressive exercise program targeting the latissimus dorsi muscle
  Arms: Combined Exercise Group (CEG); Latissimus Dorsi Exercise Group (LDEG)

SUMMARY:
The aim of this study is to investigate the effects of strengthening exercises targeting the latissimus dorsi muscle on acromiohumeral distance, shoulder function, and pain levels in individuals with rotator cuff tendinopathy. By increasing the activation of the latissimus dorsi, one of the shoulder adductor muscles, the exercises are expected to facilitate inferior gliding of the humeral head and improve subacromial distance.

Individuals aged between 18 and 50 years with a diagnosis of rotator cuff tendinopathy will be included in the study. A total of 47 participants will be enrolled and randomly assigned to one of three groups:

A group performing exercises targeting only the rotator cuff muscles, A group performing exercises targeting the latissimus dorsi muscle, A group performing a combination of both rotator cuff and latissimus dorsi exercises.

The exercise interventions will be applied over a 12-week period. Before and after the intervention, the following outcomes will be assessed:

Acromiohumeral distance (via ultrasound), Range of motion, Shoulder function and pain using the SPADI and WORC questionnaires, and Avoidance behavior using the Adap-Tr questionnaire.

DETAILED DESCRIPTION:
Subacromial pain syndrome, also referred to as rotator cuff-related shoulder pain (RCS), is characterized by pain localized to the proximal lateral aspect of the upper arm arising from the rotator cuff and other subacromial structures. Although the etiology of RCS is multifactorial, dynamic narrowing of the subacromial space due to impingement of soft tissues within this region has been proposed as a leading cause of chronic rotator cuff pathology. A lack of coordination between the rotator cuff and scapulothoracic muscles may impair shoulder neuromuscular control, leading to varying degrees of microtrauma and degenerative pathophysiological changes in the rotator cuff muscles and surrounding tissues. This dysfunction can result in further narrowing of the subacromial space. Specifically, inadequate superior rotation and posterior tilt of the scapula, combined with the inability of the rotator cuff muscles to resist the superior translation of the humeral head caused by deltoid contraction, may cause impingement of the subacromial soft tissues during overhead dynamic activities. In healthy shoulders, the acromiohumeral distance (AHD) is reported to range between 8 and 15 mm, whereas narrowing of the subacromial space (AHD < 7 mm) is considered a significant indicator of large rotator cuff tears. Moreover, in patients with rotator cuff tears, proximal migration of the humeral head is associated with tear size and decreased acromiohumeral distance.

In a young and healthy shoulder, the cranially directed forces generated during abduction are balanced by the coordinated contraction of the rotator cuff muscles. This mechanism prevents superior migration of the humerus toward the acromion and subsequent impingement of the subacromial tissues. When the contribution of the rotator cuff muscles to the abduction movement decreases, the deltoid muscle compensates for this deficit. However, this compensatory mechanism results in a force vector that is more cranially oriented rather than mediocranial. The reduction in the stabilizing force of the rotator cuff muscles may impair the ability to counteract the superior forces generated by the deltoid. Both of these changes can lead to superior migration of the humerus and pain in the subacromial tissues.

Insufficient depression of the humeral head during the abduction movement has been associated with pain patterns. During arm abduction, the rotator cuff muscles continue to be the focus of both research and clinical practice. However, several studies have demonstrated that the arm adductors-particularly the latissimus dorsi, teres major, and to a lesser extent the pectoralis major-contribute significantly to humeral head depression during abduction. Activation of these adductor muscles may reduce the mechanical load on subacromial structures during abduction. Elevation movements performed at various angles combined with adductor muscle activity may lead to a physiological increase in the subacromial space. This finding suggests the possibility of conservative treatment in patients with rotator cuff tears (RCT) by strengthening the adductor muscles.

OInvestigation of arm adductor contraction patterns during abduction has shown decreased adductor activation in individuals with rotator cuff tendinopathy. Reduced adductor activation may result in insufficient caudal forces on the humerus, leading to overload of subacromial tissues and persistence of symptoms.Therefore, adductor muscle training programs may be clinically effective in patients with rotator cuff tears. The application of neuromuscular electrical stimulation to increase activation of the teres major and pectoralis major muscles has been associated with a short-term increase in acromiohumeral distance in elderly individuals with rotator cuff tears.

The aim of this study is to increase the activation of the latissimus dorsi muscle, one of the adductor muscles, through targeted exercises, thereby increasing the acromiohumeral distance and facilitating inferior gliding of the humeral head.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 50 years
* At least 3 months of ongoing shoulder pain
* At least 3 positive tests out of 5 (Neer, Hawkins-Kennedy, Jobe, Painful Arc Sign, Pain on Resisted External Rotation)
* Ultrasound diagnosis of rotator cuff tendinopathy
* Shoulder pain during activity rated greater than 3 out of 10 on the Numeric Pain Scale
* Central Sensitization Inventory score below 40

Exclusion Criteria:

* Bilateral shoulder pain
* History of surgery or dislocation in the symptomatic shoulder
* Acromioclavicular degeneration
* Presence of shoulder capsulitis (restriction in passive glenohumeral range of motion in 2 or more directions)
* Full-thickness rotator cuff tear
* Shoulder osteoarthritis, rheumatoid arthritis, systemic inflammatory or neurological disease
* Any injection to the symptomatic shoulder within the past 6 weeks
* BMI greater than 30 kg/m2
* Refusal to participate in the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Estimated)
Dates: Start 2025-05-23 (Actual); Primary Completion 2027-05-22 (Estimated); Study Completion 2027-09-22 (Estimated)

PRIMARY OUTCOMES:
Acromio-humeral distance | Measurements will be performed at baseline and at the end of the 12th week
  The acromiohumeral distance will be assessed using ultrasonography. Measurements will be performed by a physician blinded to the participants' group assignments, ensuring assessor blinding.
  Ultrasonographic measurement of the acromiohumeral distance has been shown to be reliable (intraclass correlation coefficient > 0.90), and the minimal detectable change has been reported as 1.2 mm
Pain İntensity | Baseline and weekly up to 12 weeks
  Pain intensity will be assessed using the Visual Analog Scale (VAS) at rest, during activity, and at night. On the VAS, a score of 0 indicates no pain, while a score of 10 represents unbearable pain. Higher scores reflect greater pain intensity.he scale will be explained to the patient in a face-to-face setting, and they will be asked to mark their pain levels at rest, during activity, and at night on a 100-millimeter horizontal line.
Shoulder Range of Motion | Baseline and weekly up to 12 weeks
  ll measurements will be performed with the patient in the supine position. For shoulder flexion ROM, the patient will be asked to raise their arm upward in the sagittal plane. For shoulder abduction ROM, the patient will be instructed to move their arm laterally in the scapular plane.For external and internal rotation ROM measurements, the shoulder will be positioned at 90° of abduction and the elbow at 90° of flexion.For external rotation, the patient will be asked to move the forearm upward in the sagittal plane, with the palm facing toward themselves and in the direction of the thumb. For internal rotation, the patient will be asked to move the forearm downward in the sagittal plane, in the direction of the index finger.

SECONDARY OUTCOMES:
ADAP-Shoulder Scale (Avoidance Behavior) | Measurements will be performed at baseline and at the end of the 12th week.
  The ADAP-Shoulder Scale (Avoidance of Daily Activities due to Pain - Shoulder Scale) was developed to assess pain-related avoidance behaviors in individuals with shoulder pain (29). The ADAP-Shoulder Scale consists of 15 photographs and a questionnaire corresponding to 15 ICF activity items. It targets individuals with unilateral or bilateral shoulder pain and focuses on daily life activities while evaluating pain-related avoidance behaviors. The items are categorized into three domains: free movement (5 items), high effort (7 items), and self-care (3 items).
  Each item is rated on a scale from 0 to 10, with higher scores indicating greater avoidance behavior due to pain. The total score is calculated by multiplying the sum of the item scores by 10 and dividing by the number of items (15). The total score ranges from 0 (no avoidance) to 100 (maximum avoidance). The Turkish version of the scale has been validated (21). The minimal clinically important difference (MCID) is 5.12 points (
Shoulder Pain and Disability Index (SPADI) | At baseline and at the end of Week 12
  SPADI is a self-reported questionnaire designed to measure pain and disability associated with the shoulder. It consists of 13 items divided into two subscales: pain (5 items) and disability (8 items). Each item is scored using a visual analog scale ranging from 0 (no pain or no difficulty) to 10 (worst imaginable pain or so difficult that help is required). The total score is calculated by dividing the sum of all items by 130 and multiplying by 100. Scores range from 0 (best functional status) to 100 (worst functional status). The Turkish version of the SPADI has been validated.
Western Ontario Rotator Cuff Index (WORC) | Measurements will be performed at baseline and at the end of the 12th week.
  Western Ontario Rotator Cuff Index (WORC): The WORC is a self-assessment tool developed to measure quality of life in patients with rotator cuff pathology. It includes 21 items representing five domains that cover all aspects of health defined by the World Health Organization: physical symptoms (6 items), sports and recreation (4 items), work (4 items), lifestyle (4 items), and emotions (3 items). The total sc

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University Faculty of Physical Therapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to privacy and ethical considerations.